CLINICAL TRIAL: NCT06420284
Title: Characterization of Immunological Parameters in Different Clinical Stages of Medication-Related Osteonecrosis of the Jaw
Brief Title: Immunological Parameters Between MRONJ Stages
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist. Prof., Marmara University
Other Study IDs: MU_DHF_MI_01
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Medication-Related Osteonecrosis of Jaw

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- MRONJ Stage 0: Participants in this group are receiving antiresorptive/antiangiogenic therapy and exhibit nonspecific symptoms but no exposed bone. This stage is considered a precursor stage, where the risk of developing MRONJ is present but not yet visible through exposed bone.
- MRONJ Stage I: Individuals in this group are on antiresorptive/antiangiogenic therapy and show exposed bone without any symptoms. This stage represents the early manifestation of MRONJ, characterized by visible bone changes without associated pain or infection.
- MRONJ Stage II: This group includes patients treated with antiresorptive/antiangiogenic agents, who have exposed bone accompanied by symptoms such as pain or infection but without extensive bone involvement. This stage indicates a progression in the severity of MRONJ.
- MRONJ Stage III: Participants are undergoing antiresorptive/antiangiogenic treatment and exhibit exposed bone with symptoms, where the exposed bone extends beyond the alveolar bone, indicating advanced disease with significant bone and surrounding tissue involvement.
- At-Risk Group: This group consists of individuals receiving antiresorptive/antiangiogenic therapy who do not yet show any exposed bone or symptoms. They are considered at risk for developing MRONJ and are monitored for any potential progression.
- Healthy Control Group: This control group comprises individuals who have not received antiresorptive/antiangiogenic therapy and show no signs of exposed bone or symptoms. This group serves to provide baseline data for comparing immunological parameters against those receiving treatment.

SUMMARY:
This study aims to conduct a detailed analysis of the immunological response profiles that emerge at different clinical stages of medication-related osteonecrosis of the jaw (MRONJ). The research seeks to understand how these responses influence the pathogenesis, staging, and treatment of MRONJ. Throughout the study, cytokine levels, inflammation markers, and other immunological parameters observed at various stages will be comprehensively assessed. The results of these analyses are expected to provide insights into how stage-specific immunological variables could play a role in the diagnosis and treatment of MRONJ.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and over
* Both male and female participants
* Individuals who apply to the Oral and Maxillofacial Surgery Clinic at Marmara University Faculty of Dentistry due to medication-related osteonecrosis of the jaw during the study period
* Individuals or their legal representatives who have provided written consent to participate in the study

Exclusion Criteria:

* Non-drug-related osteonecrosis/osteomyelitis
* Osteoradionecrosis
* Metastasis to the oral region
* Individuals who have not given written consent to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population for this research comprises adults aged 18 and older, both male and female, who present with medication-related osteonecrosis of the jaw (MRONJ) at the Oral and Maxillofacial Surgery Clinic of Marmara University Faculty of Dentistry. All participants must have provided written informed consent either personally or through a legal representative to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Lymphocyte Proliferation Analysis | Baseline
  This outcome evaluates the proliferation capacity of peripheral blood mononuclear cells (PBMCs) isolated from the study participants. This analysis will help quantify and understand the dynamics of lymphocyte activation and proliferation in response to different clinical stages of MRONJ and potentially identify immunological differences that could inform therapeutic strategies.
Apoptosis Analysis in Lymphocytes | Baseline
  This outcome assesses apoptosis in lymphocytes isolated from the peripheral blood of participants included in the study. This analysis aims to quantify apoptotic processes in lymphocytes, offering insights into cell death mechanisms under varying conditions of culture and potentially relating these mechanisms to the immunopathology of MRONJ.
Cytokine Profile Analysis | Baseline
  This outcome measures the levels of specific cytokines as indicators of immunological response in MRONJ at different disease stages. The cytokines to be analyzed include IL-17, IL-2, IL-4, IL-6, IL-10, TNF-α, and IFN-γ.

CONTACTS AND LOCATIONS:
Overall Officials: Ferit Bayram, PhD, Study Chair — Marmara University Faculty of Dentistry
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruggiero SL, Dodson TB, Aghaloo T, Carlson ER, Ward BB, Kademani D. American Association of Oral and Maxillofacial Surgeons' Position Paper on Medication-Related Osteonecrosis of the Jaws-2022 Update. J Oral Maxillofac Surg. 2022 May;80(5):920-943. doi: 10.1016/j.joms.2022.02.008. Epub 2022 Feb 21. PMID 35300956